CLINICAL TRIAL: NCT03908281
Title: Exercise Training Before (Fasted) Versus After Breakfast in Type 2 Diabetes
Brief Title: Fasted Exercise Training in Type 2 Diabetes
Acronym: FED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00088195
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise; Glycated hemoglobin; Liver fat; Continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity; Fatty Liver

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: For most outcomes, including the primary outcome, the outcome assessor will be unaware of group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasted Exercise (Experimental): Exercise training will be performed in the fasted state (i.e., before breakfast).
  Interventions: Behavioral: Fasted Exercise
- Postprandial Exercise (Active Comparator): Exercise will be performed in the postprandial period (i.e., after breakfast)
  Interventions: Behavioral: Postprandial Exercise

INTERVENTIONS:
Behavioral: Fasted Exercise — Exercise training will take place 3 times per week and will progress to 60 minutes at a workload corresponding to 80% of Ventilatory Threshold.
  Arms: Fasted Exercise
Behavioral: Postprandial Exercise — Exercise training will take place 3 times per week and will progress to 60 minutes at a workload corresponding to 80% of Ventilatory Threshold.
  Arms: Postprandial Exercise

SUMMARY:
This study compares aerobic exercise training performed before breakfast (i.e., in the fasted state) to similar training performed after breakfast in people with type 2 diabetes. Training will take place over 16 weeks.

DETAILED DESCRIPTION:
People with type 2 diabetes (T2D) are encouraged to increase their physical activity (PA). Sometimes, increasing the amount of PA can be difficult. Therefore, simply recommending that individuals preform more exercise may not be effective in the long term. Recent short-term studies have started to explore how to maximize the effect of a single bout of exercise. For example, short term studies suggest that exercise performed after a meal may decrease blood sugars more than exercise performed after a meal. However, research in people without diabetes shows this may not be the best approach in the long-term. To date, no long-term study has compared the effects of exercise performed at different times of the day in people with T2D.

This study will compare the effects of 16 weeks of regular exercise before breakfast compared to 16 weeks of regular exercise after breakfast. It is expected that exercise before breakfast (i.e., in the fasted state) will lead to greater improvements in blood sugar control, without the addition of more exercise. It could be very motivating for people with diabetes to know that they can get more benefits from exercise by changing when exercise is performed, rather than trying to increase the amount of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosed type 2 diabetes
* Treated with diet and/or glucose lowering medications, but not insulin, for at least 6 months
* Sedentary (defined as reaching <150 minutes of aerobic exercise per week)
* A1C below 9.0%
* BMI ≥25 kg/m2
* Central obesity as determined by waist circumference according to Diabetes Canada cutoffs:
* greater or equal to 94cm for males of European, Sub-Saharan African, Eastern Mediterranean and Middle Eastern descent,
* greater or equal to 90cm for males of South Asian, Chinese, Japanese, South and Central American descent,
* greater or equal to 80cm for females
* Able to walk for 50 minutes

Exclusion Criteria:

* Smoking
* Consuming more than 10 alcoholic drinks/week
* History of stroke, myocardial infarction, or coronary artery disease
* Resting heart rate <100 bpm
* Resting blood pressure <160/100 mmHg
* Implantable device, such as a pacemaker, that would not be safe for Magnetic Resonance Imaging

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Concentration of HbA1c (mmol/mol) | Change from baseline HbA1c at 16 weeks
  Glycated Hemoglobin
Liver fat (%) | Change from baseline liver fat at 16 weeks
  Intra-hepatic fat measured by Magnetic Resonance Imaging

SECONDARY OUTCOMES:
Pancreatic fat (%) | Change from pancreatic fat at 16 weeks
  Pancreatic fat measured by Magnetic Resonance Imaging
Muscle fat (%) | Change from baseline muscle fat at 16 weeks
  Muscle fat measured by Magnetic Resonance Imaging
Concentrations of Fasting glucose | Change from baseline fasting glucose at 16 weeks
  Plasma glucose measured after an overnight fast
Concentrations of Fasting insulin | Change from baseline fasting insulin at 16 weeks
  Plasma insulin measured after an overnight fast
Concentrations of Fasting lipids | Change from baseline fasting lipids at 16 weeks
  Plasma total cholesterol, HDL-Cholesterol, LDL-Cholesterol and Triglycerides measured after an overnight fast
Concentrations of Liver enzymes | Change from baseline liver enzymes at 16 weeks
  Alanine aminotransferase, Aspartate aminotransferase measured after an overnight fast
Aerobic fitness | Change from baseline aerobic fitness at 16 weeks
  Submaximal exercise test to determine ventilatory threshold
Height (centimeters) | Change from baseline height at 16 weeks
  Standing height
Waist circumference (centimeters) | Change from baseline waist circumference at 16 weeks
  Waist circumference (between 12 rib and iliac crest) measures in centimeters
Hip circumference (centimeters) | Change from baseline hip circumference at 16 weeks
  Hip circumference (between 12 rib and iliac crest) measures in centimeters
Body weight (kilograms) | Change from baseline weight at 16 weeks
  Weight will be measured in kilograms
Continuous glucose monitoring | Change from the first two to the last two weeks of the 16 week interventions
  Continuous glucose monitoring outcomes (e.g., 24-hour mean glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Normand Boulé, PhD, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
We plan to share all of the data related to study outcomes pm am open access website through the University of Alberta "Education and Research Archive" (ERA). Individual participant characteristics that could be used to identify participants (age, sex, height, weight) will not be be placed on ERA.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will become available one year after the completion of the trial.
Access Criteria: The outcome data will be open access through the University of Alberta "Education and Research Archive" (ERA) website. Other participant characteristics will be available as meta-data.
URL: https://era.library.ualberta.ca

REFERENCES:
- [Derived] Rees JL, Walesiak D, Thompson R, Mager D, Senior P, Boule NG. HbA1c and Liver Fat After 16 Weeks of Fasted versus Fed Exercise Training in Adults With Type 2 Diabetes. Med Sci Sports Exerc. 2025 Jan 1;57(1):106-114. doi: 10.1249/MSS.0000000000003552. Epub 2024 Sep 16. PMID 39283231